CLINICAL TRIAL: NCT01506271
Title: A Phase II, Randomized, Active Comparator-Controlled Clinical Trial to Study the Safety, Tolerability, and Efficacy of MK-7655 + Imipenem/Cilastatin Versus Imipenem/Cilastatin Alone in Patients With Complicated Intra-Abdominal Infection [cIAI]
Brief Title: Study of the Safety, Tolerability, and Efficacy of Relebactam (MK-7655) + Imipenem/Cilastatin Versus Imipenem/Cilastatin Alone to Treat Complicated Intra-Abdominal Infection [cIAI] (MK-7655-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7655-004; 2011-005686-20 (EudraCT Number); MK-7655-004 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Intra-abdominal Infections
Keywords: Complicated Intra-abdominal Infections
MeSH Terms: conditions — Intraabdominal Infections | interventions — relebactam; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Relebactam 250 mg with imipenem/cilastatin (Experimental): Participants randomized to receive relebactam 250 mg will be administered 250 mg doses of relebactam IV in a blinded fashion once every 6 hours with each dose infused over a 30-minute interval. A 500 mg dose of imipenem/cilastatin will be administered in an open-label fashion once every 6 hours with each dose infused over a 30-minute interval.
  Interventions: Drug: Relebactam 250 mg; Drug: Imipenem/cilastatin
- Relebactam 125 mg with imipenem/cilastatin (Experimental): Participants randomized to receive relebactam 125 mg will be administered 125 mg doses of relebactam IV, in a blinded-treatment fashion once every 6 hours with each dose infused over a 30-minute interval. A 500 mg dose of imipenem/cilastatin will be administered IV in an open-label fashion once every 6 hours with each dose infused over a 30-minute interval.
  Interventions: Drug: Relebactam 125 mg; Drug: Imipenem/cilastatin
- Placebo to relebactam with imipenem/cilastatin (Placebo Comparator): Participants randomized to receive placebo for relebactam will receive a placebo-matching infusion of IV normal saline (0.9%) once every 6 hours. A 500 mg dose of imipenem/cilastatin will be administered IV in an open-label fashion once every 6 hours with each dose infused over a 30-minute interval.
  Interventions: Drug: Imipenem/cilastatin; Drug: Matching placebo to relebactam

INTERVENTIONS:
Drug: Relebactam 250 mg — Relebactam 250 mg IV every 6 hours for a minimum of 96 hours
  Other Names: MK-7655
  Arms: Relebactam 250 mg with imipenem/cilastatin
Drug: Relebactam 125 mg — Relebactam 125 mg IV every 6 hours for a minimum of 96 hours
  Other Names: MK-7655
  Arms: Relebactam 125 mg with imipenem/cilastatin
Drug: Imipenem/cilastatin — A 500 mg dose of imipenem/cilastatin will be administered IV in an open-label fashion once every 6 hours with each dose infused over a 30-minute interval.
Drug: Matching placebo to relebactam — Placebo-matching infusion of IV normal saline (0.9%) once every 6 hours.
  Arms: Placebo to relebactam with imipenem/cilastatin

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of adding 125 mg or 250 mg doses of relebactam (MK-7655) to imipenem/cilastatin in adults 18 years or older with Complicated Intra-Abdominal Infection (cIAI). The primary hypothesis is that the relebactam + imipenem/cilastatin treatment regimen is non-inferior to treatment with imipenem/cilastatin alone with respect to the percentage of participants with a favorable clinical response at completion of intravenous (IV) study therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected and/or bacteriologically documented cIAI requiring hospitalization and treatment with IV antibiotic therapy.
* Enrolled intraoperatively or postoperatively on the basis of operative findings OR enrolled preoperatively on the basis of compelling preoperative clinical findings.

Exclusion Criteria:

* Infection which should be managed by Staged Abdominal Repair (STAR) or open abdomen technique.
* Acute Physiology and Chronic Health Evaluation II (APACHE II) score greater than 30.
* Any amount of effective antibiotic therapy after obtaining the culture for admission to this study and prior to the administration of the first dose of IV study therapy.
* An infection which has been treated with >24 hours of systemic antibiotic therapy known to be effective against the presumed or documented etiologic pathogen(s) within the 72-hour period immediately prior to consideration for entry into the study.
* History of serious allergy, hypersensitivity (e.g., anaphylaxis), or any serious reaction to carbapenem antibiotics, any cephalosporins, penicillins, or other β-lactam agents.
* History of serious allergy, hypersensitivity (e.g., anaphylaxis), or any serious reaction to other β-lactamase inhibitors (e.g., tazobactam, sulbactam, clavulanic acid).
* History of a seizure disorder (requiring ongoing treatment with anticonvulsive therapy or prior treatment with anti-convulsive therapy in the last 3 years).
* Currently being treated with valproic acid or has used valproic acid in the 2 weeks prior to screening.
* Rapidly progressive or terminal illness (unlikely to survive the approximately 6- to 8-week study period).
* Pregnant or expecting to conceive, breastfeeding, or plans to breast feed within 1 month of completion of the study.
* Participant in whom a response to IV study therapy within the timeframe of treatment specified in this protocol is considered unlikely.
* Concurrent infection that would interfere with evaluation of response to the study antibiotics.
* Need for concomitant systemic antimicrobial agents in addition to those designated in the various study treatment groups.
* cIAI due to a confirmed fungal pathogen.
* Currently receiving immunosuppressive therapy, including use of high-dose corticosteroids.
* Prior recipient of a renal transplantation.
* Estimated or actual creatinine clearance of <50 mL/minute.
* History of any other illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering the study drug to the patient.
* Laboratory abnormalities as specified in protocol.
* Currently participating in, or has participated in any other clinical study involving the administration of investigational or experimental medication (not licensed by regulatory agencies) at the time of presentation or during the previous 30 days prior to screening or is anticipated to participate in such a clinical study during the course of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2014-08-12 (Actual); Study Completion 2014-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lucasti C, Vasile L, Sandesc D, Venskutonis D, McLeroth P, Lala M, Rizk ML, Brown ML, Losada MC, Pedley A, Kartsonis NA, Paschke A. Phase 2, Dose-Ranging Study of Relebactam with Imipenem-Cilastatin in Subjects with Complicated Intra-abdominal Infection. Antimicrob Agents Chemother. 2016 Sep 23;60(10):6234-43. doi: 10.1128/AAC.00633-16. Print 2016 Oct. PMID 27503659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults 18 years or older with complicated intra-abdominal infection (cIAI) requiring treatment with intravenous (IV) antibiotic therapy were enrolled in this study.
Groups:
- Relebactam 250 mg With Imipenem/Cilastatin: Participants received relebactam 250 mg IV with imipenem/cilastatin 500 mg IV every 6 hours for a minimum of 96 hours
- Relebactam 125 mg With Imipenem/Cilastatin: Participants received relebactam 125 mg IV with imipenem/cilastatin 500 mg IV every 6 hours for a minimum of 96 hours
- Placebo to Relebactam With Imipenem/Cilastatin: Participants received matching placebo to relebactam (normal saline 0.9%) IV with imipenem/cilastatin 500 mg IV every 6 hours for a minimum of 96 hours
Period: Overall Study
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Started | 118 | 116 | 117
Treated | 117 | 116 | 114
Completed | 114 | 109 | 114
Not Completed | 4 | 7 | 3
Not completed — Progressive disease | 0 | 1 | 0
Not completed — Protocol Violation | 3 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Insufficient supply of study drug | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin | Total
Number analyzed (Participants) | 118 | 116 | 117 | 351
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.3 (18.9) | 49.8 (17.4) | 49.1 (17.8) | 49.1 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 54 | 51 | 149
  Male | 74 | 62 | 66 | 202

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Favorable Clinical Response at Completion of IV Study Therapy
Description: A favorable clinical response was assessed by the clinical investigator as a cure, and was defined as a situation where all or most pre-therapy signs and symptoms of the index infection had resolved, or returned to pre-infection status, and no additional antibiotic therapy was required.
Time Frame: 4 to 14 days post initiation of intravenous (IV) study therapy (up to postrandomization Day 14)
Population: Those who had cIAI; a culture from the infection that grew one Gram negative pathogen; no protocol deviations; received ≥ 96 hours of IV therapy. Two participants treated with relebactam 250 mg, one with relebactam 125 mg, and two with placebo, all with indeterminate or missing responses, were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 81 | 86 | 83
Percentage of participants | 96.3 [89.6 to 99.2] | 98.8 [93.7 to 100] | 95.2 [88.1 to 98.7]
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; MK-7655 250 mg - Placebo: Percentage Difference; Test type: Non-Inferiority — Non-inferiority test based on unconditional asymptotic Miettinen and Nurminen method without stratification; p < 0.001, Miettinen and Nurminen; Percentage Difference = 1.1, 95% CI 2-sided [-6.2 to 8.6] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Non-Inferiority — Non-inferiority test based on unconditional asymptotic Miettinen and Nurminen method without stratification; p < 0.001, Miettinen and Nurminen; Percentage Difference = 3.7, 95% CI 2-sided [-2.0 to 10.8] — Relebactam minus Placebo

2. Primary Outcome: Percentage of Participants With an Elevated Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) Laboratory Values That Are Greater Than or Equal to 5X the Upper Limit of Normal (ULN)
Description: Pre-specified events of interest were confirmed (i.e., verified by repeat testing) elevated AST or ALT laboratory value that is greater than or equal to 5 X ULN as a result of within-protocol-specific testing or unscheduled testing.
Time Frame: Up to 14 days following completion of all study therapy (up to Day 28)
Population: All randomized participants who received at least one dose of IV study therapy, based on the therapy they actually received
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 117 | 116 | 114
Percentage of participants | 1.7 | 0 | 1.8
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Other — Test for a non-zero difference; p = 0.979, Miettinen and Nurminen; Percentage Difference = 0, 95% CI 2-sided [-4.7 to 4.5] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Other — Test for a non-zero difference; p = 0.153, Miettinen and Nurminen; Percentage Difference = -1.8, 95% CI 2-sided [-6.2 to 1.5] — Relebactam minus Placebo

3. Primary Outcome: Percentage of Participants With Elevated AST or ALT Laboratory Values >= 3X the ULN, Total Bilirubin >= 2X the ULN, and Alkaline Phosphatase Values < 2X the ULN
Description: Pre-specified events of interest were a confirmed (i.e., verified by repeat testing) elevated AST or ALT laboratory value that is greater than or equal to 3X ULN, as well as elevated total bilirubin greater than or equal to 2X the ULN, and alkaline phosphatase values that are less than 2X the ULN, as a result of within-protocol-specific testing or unscheduled testing.
Time Frame: Up to 14 days following completion of all study therapy (up to Day 28)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 117 | 116 | 114
Percentage of participants | 0.9 | 0 | 0
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Other — Test for a non-zero difference; p = 0.324, Miettinen and Nurminen; Percentage Difference = 0.9, 95% CI 2-sided [-2.4 to 4.7] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Other — Test for a non-zero difference; p > 0.999, Miettinen and Nurminen; Percentage Difference = 0, 95% CI 2-sided [-3.3 to 3.2] — Relebactam minus Placebo

4. Primary Outcome: Percentage of Participants With Any Adverse Event (AE)
Description: An adverse event (AE) is any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the medicinal product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the medicinal product, is also an AE.
Time Frame: Up to 14 days following completion of all study therapy (up to Day 28)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 117 | 116 | 114
Percentage of participants | 48.7 | 47.4 | 41.2
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 7.5, 95% CI 2-sided [-5.4 to 20.1] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 6.2, 95% CI 2-sided [-6.7 to 18.8] — Relebactam minus Placebo

5. Primary Outcome: Percentage of Participants With Any Serious Adverse Event (SAE)
Description: A serious adverse event (SAE) is any AE occurring at any dose that is life threatening; results in a persistent or significant disability/incapacity; prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; or results in death.
Time Frame: Up to 14 days following completion of all study therapy (up to Day 28)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 117 | 116 | 114
Percentage of participants | 3.4 | 9.5 | 7
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -3.6, 95% CI 2-sided [-10.3 to 2.4] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 2.5, 95% CI 2-sided [-5.0 to 10.1] — Relebactam minus Placebo

6. Primary Outcome: Percentage of Participants With Any Drug-related AE
Description: An AE is any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the medicinal product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the medicinal product, is also an AE. A drug-related AE is a AE determined by the investigator to be possibly, probably or definitely related to drug treatment.
Time Frame: Up to 14 days following completion of all study therapy (up to Day 28)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 117 | 116 | 114
Percentage of participants | 13.7 | 13.8 | 9.6
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 4.0, 95% CI 2-sided [-4.5 to 12.7] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 4.1, 95% CI 2-sided [-4.4 to 12.8] — Relebactam minus Placebo

7. Primary Outcome: Percentage of Participants With Any Drug-related SAE
Description: A SAE is any AE occurring at any dose that is life threatening; results in a persistent or significant disability/incapacity; prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; or results in death. A drug-related SAE is a SAE determined by the investigator to be possibly, probably or definitely related to drug treatment.
Time Frame: Up to 42 days following completion of all study therapy (up to Day 56)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 117 | 116 | 114
Percentage of participants | 0.9 | 0 | 0.9
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 0, 95% CI 2-sided [-4.0 to 3.9] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -0.9, 95% CI 2-sided [-4.8 to 2.4] — Relebactam minus Placebo

8. Primary Outcome: Percentage of Participants Who Discontinued IV Study Therapy Due to an AE
Description: An AE is any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the medicinal product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the medicinal product, is also an AE. AEs assessed by the investigator that caused discontinuation of participant treatment are presented.
Time Frame: Up to 14 days post initiation of IV study therapy (up to 14 days)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 117 | 116 | 114
Percentage of participants | 0.9 | 4.3 | 2.6
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -1.8, 95% CI 2-sided [-6.7 to 2.3] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 1.7, 95% CI 2-sided [-3.7 to 7.4] — Relebactam minus Placebo

9. Primary Outcome: Percentage of Participants Who Discontinued IV Study Therapy Due to a Drug-related AE
Description: An AE is any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the medicinal product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the medicinal product, is also an AE. A drug-related AE is an AE determined by the investigator to be possibly, probably or definitely related to drug treatment. Drug-related AEs assessed by the investigator that caused discontinuation of participant treatment are presented.
Time Frame: Up to 14 days post initiation of IV study therapy (up to 14 days)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 117 | 116 | 114
Percentage of participants | 0 | 0.9 | 2.6
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -2.6, 95% CI 2-sided [-7.5 to 0.6] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -1.8, 95% CI 2-sided [-6.7 to 2.4] — Relebactam minus Placebo

10. Primary Outcome: Percentage of Participants With Specific AEs With Incidence of >= 4 Participants in One Treatment Group
Description: An AE is any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the medicinal product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the medicinal product, is also an AE. AE preferred terms, with incidence greater than or equal to 4 in one treatment group are presented. AEs preferred terms which did not achieve this threshold are not reported. AE preferred terms are based on MedDRA version 17.0.
Time Frame: Up to 42 days following completion of all study therapy (up to Day 56)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 117 | 116 | 114
Percentage of participants
  Diarrhoea | 6.0 | 6.0 | 4.4
  Nausea | 6.8 | 7.8 | 7.0
  Vomiting | 6.0 | 7.8 | 2.6
  Post-operative wound infection | 2.6 | 1.7 | 4.4
  Seroma | 0.9 | 4.3 | 0
  ALT increased | 4.3 | 4.3 | 3.5
  AST increased | 4.3 | 4.3 | 2.6
  Lipase increased | 2.6 | 1.7 | 3.5
  Hypertension | 0 | 2.6 | 3.5
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Diarrhoea; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 1.6, 95% CI 2-sided [-4.7 to 8.1] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Diarrhoea; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 1.6, 95% CI 2-sided [-4.6 to 8.2] — Relebactam minus Placebo
Statistical Analysis 3: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Nausea; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -0.2, 95% CI 2-sided [-7.3 to 6.9] — Relebactam minus Placebo
Statistical Analysis 4: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Nausea; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 0.7, 95% CI 2-sided [-6.5 to 8.0] — Relebactam minus Placebo
Statistical Analysis 5: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Vomiting; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 3.4, 95% CI 2-sided [-2.3 to 9.6] — Relebactam minus Placebo
Statistical Analysis 6: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Vomiting; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 5.1, 95% CI 2-sided [-0.7 to 11.8] — Relebactam minus Placebo
Statistical Analysis 7: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Postoperative Infection; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -1.8, 95% CI 2-sided [-7.6 to 3.5] — Relebactam minus Placebo
Statistical Analysis 8: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Postoperative Infection; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -2.7, 95% CI 2-sided [-8.4 to 2.2] — Relebactam minus Placebo
Statistical Analysis 9: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Seroma; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 0.9, 95% CI 2-sided [-2.4 to 4.7] — Relebactam minus Placebo
Statistical Analysis 10: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Seroma; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 4.3, 95% CI 2-sided [1.0 to 9.7] — Relebactam minus Placebo
Statistical Analysis 11: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - ALT increased; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 0.8, 95% CI 2-sided [-5.0 to 6.6] — Relebactam minus Placebo
Statistical Analysis 12: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - ALT increased; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 0.8, 95% CI 2-sided [-4.9 to 6.7] — Relebactam minus Placebo
Statistical Analysis 13: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - AST increased; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 1.6, 95% CI 2-sided [-3.7 to 7.3] — Relebactam minus Placebo
Statistical Analysis 14: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - AST increased; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 1.7, 95% CI 2-sided [-3.7 to 7.4] — Relebactam minus Placebo
Statistical Analysis 15: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Lipase increased; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -0.9, 95% CI 2-sided [-6.5 to 4.2] — Relebactam minus Placebo
Statistical Analysis 16: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Lipase increased; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -1.8, 95% CI 2-sided [-7.2 to 3.0] — Relebactam minus Placebo
Statistical Analysis 17: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Relebactam 125 mg With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Hypertension; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -3.5, 95% CI 2-sided [-8.7 to -0.3] — Relebactam minus Placebo
Statistical Analysis 18: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Hypertension; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -0.9, 95% CI 2-sided [-6.4 to 4.3] — Relebactam minus Placebo

11. Secondary Outcome: Percentage of Participants With a Favorable Clinical Response at Completion of IV Study Therapy in Participants Who Have Imipenem-resistant, Gram-negative cIAI Infections.
Description: A favorable clinical response is assessed by the clinical investigator as a cure, and is defined as a situation where all or most pre-therapy signs and symptoms of the index infection have resolved, or returned to pre-infection status, and no additional antibiotic therapy is required.
Time Frame: 4 to 14 days post initiation of IV study therapy (up to postrandomization day 14).
Population: Met the protocol definition of cIAI; had a culture from the site of infection, that grew Gram-negative pathogen; had no significant deviations from the protocol that could impact the efficacy assessment; received ≥ 96 hours of IV study therapy; and had imipenem-resistant, gram negative cIAI infections.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 14 | 9 | 11
Percentage of participants | 100 [76.8 to 100] | 100 [66.4 to 100] | 100 [71.5 to 100]
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Superiority; p > 0.999, Fisher Exact; Percentage Difference = 0, 95% CI 2-sided [0 to 0] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Superiority; p > 0.999, Fisher Exact; Percentage Difference = 0, 95% CI 2-sided [0 to 0] — Relebactam minus Placebo

12. Secondary Outcome: Percentage of Participants With a Favorable Clinical Response at Early Follow-up
Description: as for outcome 11
Time Frame: Up to 9 days following completion of all study therapy (up to Day 23)
Population: Met the protocol definition of cIAI; had a culture from the site of infection, that grew Gram-negative pathogen; had no significant deviations from the protocol that could impact the efficacy assessment; received ≥ 96 hours of IV study therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 79 | 86 | 81
Percentage of participants | 94.9 [87.5 to 98.6] | 94.2 [87.0 to 98.1] | 96.3 [89.6 to 99.2]
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Non-Inferiority — Unconditional asymptotic Miettinen and Nurminen method without stratification; p = 0.001, Miettinen and Nurminen; Percentage Difference = -1.4, 95% CI 2-sided [-9.1 to 6.0] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Non-Inferiority — Unconditional asymptotic Miettinen and Nurminen method without stratification; p = 0.002, Miettinen and Nurminen; Percentage Difference = -2.1, 95% CI 2-sided [-9.7 to 5.3] — Relebactam minus Placebo

13. Secondary Outcome: Percentage of Participants With a Favorable Microbiological Response at Completion of IV Study Therapy
Description: A favorable microbiological response is assessed by the clinical investigator, and is defined as the eradication or presumptive eradication of all bacterial pathogens identified at baseline.
Time Frame: Up to 14 days post initiation of IV study therapy (up to postrandomization day 14)
Population: Met the protocol definition of cIAI; had a pre-study/post operative culture from the site of infection grew at least one Gram-negative enteric and/or anaerobic pathogen; had no significant deviations from the protocol that could impact the efficacy assessment; and received ≥ 96 hours of IV study therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 83 | 86 | 84
Percentage of participants | 97.6 [91.6 to 99.7] | 100 [95.8 to 100] | 97.6 [91.7 to 99.7]
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Non-Inferiority — Two participants with indeterminate or missing response were excluded from the analysis; p < 0.001, Miettinen and Nurminen; Percentage Difference = 0, 95% CI 2-sided [-6.3 to 6.2] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Non-Inferiority — Two participants with indeterminate or missing response were excluded from the analysis; p < 0.001, Miettinen and Nurminen; Percentage Difference = 2.4, 95% CI 2-sided [-2.0 to 8.3] — Relebactam minus Placebo

14. Secondary Outcome: Percentage of Participants With a Favorable Microbiological Response at Early Follow-up
Description: as for outcome 13
Time Frame: Up to 9 days following completion of all study therapy (up to Day 23)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 78 | 82 | 80
Percentage of participants | 97.4 [91.0 to 99.7] | 97.6 [91.5 to 99.7] | 97.5 [91.3 to 99.7]
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Non-Inferiority — Eight participants with indeterminate or missing response were excluded from the analysis; p < 0.001, Miettinen and Nurminen; Percentage Difference = -0.1, 95% CI 2-sided [-6.7 to 6.4] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Non-Inferiority — Eight participants with indeterminate or missing response were excluded from the analysis; p < 0.001, Miettinen and Nurminen; Percentage Difference = 0.1, 95% CI 2-sided [-6.3 to 6.5] — Relebactam minus Placebo

15. Secondary Outcome: Percentage of Participants With a Favorable Clinical Response at Late Follow-up
Description: as for outcome 11
Time Frame: Up to 42 days following completion of all study therapy (up to Day 56)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 79 | 85 | 79
Percentage of participants | 93.7 [85.8 to 97.9] | 95.3 [88.4 to 98.7] | 94.9 [87.5 to 98.6]
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Non-Inferiority — Non-inferiority test based on Unconditional asymptotic Miettinen and Nurminen method without stratification; p = 0.002, Miettinen and Nurminen; Percentage Difference = -1.3, 95% CI 2-sided [-9.6 to 6.9] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Non-Inferiority — Unconditional asymptotic Miettinen and Nurminen method without stratification; p < 0.001, Miettinen and Nurminen; Percentage Difference = 0.4, 95% CI 2-sided [-7.2 to 8.2] — Relebactam minus Placebo

16. Secondary Outcome: Percentage of Participants With a Favorable Microbiological Response at Late Follow-up
Description: as for outcome 13
Time Frame: Up to 42 days following completion of all study therapy (up to Day 56)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 78 | 81 | 78
Percentage of participants | 96.2 [89.2 to 99.2] | 97.5 [91.4 to 99.7] | 96.2 [89.2 to 99.2]
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference; Test type: Non-Inferiority — Eight participants with indeterminate or missing response were excluded from the analysis; p < 0.001, Miettinen and Nurminen; Percentage Difference = 0, 95% CI 2-sided [-7.4 to 7.4] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference; Test type: Non-Inferiority — Eight participants with indeterminate or missing response were excluded from the analysis; p < 0.001, Miettinen and Nurminen; Percentage Difference = 1.4, 95% CI 2-sided [-5.2 to 8.6] — Relebactam minus Placebo

17. Primary Outcome: Percentage of Participants With Predefined Limit of Change (PDLC) With Incidence of >= 4 Participants in One Treatment Group
Description: Predefined limit of change (PDLC) are presented based on values from the following laboratory tests on serum: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (Bil), and alkaline phosphatase (AP). Results are presented for PDLC from tests with reported incidence greater than or equal to 4 participants in one treatment group. Laboratory tests which did not achieve the PDLC threshold are not reported.
Time Frame: Up to 42 days following completion of all study therapy (up to Day 56)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 117 | 116 | 114
Percentage of participants
  ALT >2.5-5.0 X Baseline | 3.6 | 2.6 | 9.1
  ALT >5.0 X Baseline | 4.5 | 6.1 | 3.6
  AST >2.5-5.0 X Baseline | 14.5 | 14.0 | 9.2
  AP >2.5-5.0 X Baseline | 6.3 | 2.6 | 5.5

18. Primary Outcome: Percentage of Participants With System Organ Class (SOC) With AEs With Incidence of >= 4 Participants in One Treatment Group
Description: A system organ class (SOC) is the highest level of terminology used to describe disorders of the human body, and distinguishes by either anatomical or physiological systems, disease origin or purpose. SOCs with AE incidence greater than or equal to 4 in one treatment group are presented. SOCs with AE incidence which did not achieve this threshold are not reported. SOCs are based on MedDRA version 17.0.
Time Frame: Up to 42 days following completion of all study therapy (up to Day 56)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
Number analyzed (Participants) | 117 | 116 | 114
Percentage of participants
  Blood and lymphatic system disorders | 4.3 | 0.9 | 5.3
  Cardiac disorders | 2.6 | 3.4 | 2.6
  Gastrointestinal disorders | 18.8 | 17.2 | 13.2
  General disorders admin. site conditions | 7.7 | 5.2 | 3.5
  Infections and infestations | 11.1 | 7.8 | 7.0
  Injury, poisoning, procedural complications | 4.3 | 6.9 | 5.3
  Investigations | 11.1 | 10.3 | 12.3
  Nervous system disorders | 1.7 | 3.4 | 4.4
  Psychiatric disorders | 3.4 | 3.4 | 3.5
  Renal and urinary disorders | 1.7 | 1.7 | 3.5
  Respiratory, thoracic, mediastinal disorders | 1.7 | 4.3 | 6.1
  Skin, subcutaneous tissue disorders | 4.3 | 1.7 | 1.8
  Vascular disorders | 2.6 | 6.0 | 6.1
Statistical Analysis 1: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Blood, lymphatic; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -1.0, 95% CI 2-sided [-7.3 to 5.1] — Relebactam minus Placebo
Statistical Analysis 2: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Blood, lymphatic; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -4.4, 95% CI 2-sided [-10.3 to 0.1] — Relebactam minus Placebo
Statistical Analysis 3: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Cardiac disorder; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -1.0, 95% CI 2-sided [-5.2 to 5.0] — Relebactam minus Placebo
Statistical Analysis 4: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Cardiac disorder; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 0.8, 95% CI 2-sided [-4.5 to 6.3] — Relebactam minus Placebo
Statistical Analysis 5: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - GI disorders; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 5.6, 95% CI 2-sided [-3.9 to 15.3] — Relebactam minus Placebo
Statistical Analysis 6: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - GI disorders; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 4.1, 95% CI 2-sided [-5.4 to 13.6] — Relebactam minus Placebo
Statistical Analysis 7: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Gen. dis & admin; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 4.2, 95% CI 2-sided [-2.0 to 11.0] — Relebactam minus Placebo
Statistical Analysis 8: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Gen. dis & admin; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 1.7, 95% CI 2-sided [-4.2 to 7.8] — Relebactam minus Placebo
Statistical Analysis 9: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Infect. & Infest; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 4.1, 95% CI 2-sided [-3.6 to 12.0] — Relebactam minus Placebo
Statistical Analysis 10: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Infect. & Infest; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 0.7, 95% CI 2-sided [-6.5 to 8.0] — Relebactam minus Placebo
Statistical Analysis 11: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Injury, poison; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -1.0, 95% CI 2-sided [-7.3 to 5.1] — Relebactam minus Placebo
Statistical Analysis 12: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 1250mg - Placebo: Percentage Difference - Injury, poison; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 1.6, 95% CI 2-sided [-5.0 to 8.5] — Relebactam minus Placebo
Statistical Analysis 13: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Investigations; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -1.2, 95% CI 2-sided [-9.8 to 7.4] — Relebactam minus Placebo
Statistical Analysis 14: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Investigations; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -1.9, 95% CI 2-sided [-10.5 to 6.5] — Relebactam minus Placebo
Statistical Analysis 15: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Nervous System; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -2.7, 95% CI 2-sided [-8.4 to 2.2] — Relebactam minus Placebo
Statistical Analysis 16: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Nervous System; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -2.7, 95% CI 2-sided [-8.4 to 2.2] — Relebactam minus Placebo
Statistical Analysis 17: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Psychiatric disorders; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -0.1, 95% CI 2-sided [-5.7 to 5.4] — Relebactam minus Placebo
Statistical Analysis 18: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Psychiatric disorders; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -0.1, 95% CI 2-sided [-5.7 to 5.5] — Relebactam minus Placebo
Statistical Analysis 19: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Renal & Urinary; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -1.8, 95% CI 2-sided [-7.2 to 3.0] — Relebactam minus Placebo
Statistical Analysis 20: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Renal & Urinary; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -1.8, 95% CI 2-sided [-7.2 to 3.0] — Relebactam minus Placebo
Statistical Analysis 21: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Resp. & chest; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -4.4, 95% CI 2-sided [-10.7 to 0.7] — Relebactam minus Placebo
Statistical Analysis 22: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Resp. & chest; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -1.8, 95% CI 2-sided [-8.4 to 4.4] — Relebactam minus Placebo
Statistical Analysis 23: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Skin & subcutan; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 2.5, 95% CI 2-sided [-2.4 to 8.1] — Relebactam minus Placebo
Statistical Analysis 24: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Skin & subcutan; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = 0, 95% CI 2-sided [-4.7 to 4.5] — Relebactam minus Placebo
Statistical Analysis 25: Comparison: Relebactam 250 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 250 mg - Placebo: Percentage Difference - Vascular disorders; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -3.6, 95% CI 2-sided [-9.9 to 2.0] — Relebactam minus Placebo
Statistical Analysis 26: Comparison: Relebactam 125 mg With Imipenem/Cilastatin vs Placebo to Relebactam With Imipenem/Cilastatin; Relebactam 125 mg - Placebo: Percentage Difference - Vascular disorders; Test type: Other — Unconditional asymptotic Miettinen and Nurminen method without stratification; Percentage Difference = -0.1, 95% CI 2-sided [-6.9 to 6.6] — Relebactam minus Placebo

ADVERSE EVENTS:
Time Frame: During study therapy and the protocol-specified follow-up period following end of study therapy (up to 28 days for non-serious AEs and up to 56 days for serious AEs)
Description: Population analyzed is all randomized participants who received at least one dose of IV study therapy. Participants with All-Cause Mortality were determined by the investigator to include some participants discontinued due to an adverse event, and progressive disease.
Arm/Group | Relebactam 250 mg With Imipenem/Cilastatin | Relebactam 125 mg With Imipenem/Cilastatin | Placebo to Relebactam With Imipenem/Cilastatin
All-Cause Mortality (participants affected / at risk) | 0/117 | 3/116 | 0/114
Serious Adverse Events (participants affected / at risk) | 4/117 | 13/116 | 8/114
Other Adverse Events (participants affected / at risk) | 16/117 | 15/116 | 13/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relebactam 250 mg With Imipenem/Cilastatin (N=117) | Relebactam 125 mg With Imipenem/Cilastatin (N=116) | Placebo to Relebactam With Imipenem/Cilastatin (N=114)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relebactam 250 mg With Imipenem/Cilastatin (N=117) | Relebactam 125 mg With Imipenem/Cilastatin (N=116) | Placebo to Relebactam With Imipenem/Cilastatin (N=114)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 6 (6) | 5 (5)
Nausea (Gastrointestinal disorders) | 8 (9) | 9 (9) | 8 (9)
Vomiting (Gastrointestinal disorders) | 7 (7) | 9 (9) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.